CLINICAL TRIAL: NCT03801200
Title: A Prospective, Multicenter, Randomized Controlled Trial of Apatinib Combined With Radiotherapy in Patient With Brain Metastases From Drive Gene Negative NSCLC
Brief Title: Apatinib Combined With Radiotherapy in Patient With BM From Drive Gene Negative NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, HAN GUANG, Radiation Oncologist, Hubei Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBCH RT-2019-01
Record Dates: First submitted 2018-12-30; First posted 2019-01-11 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: NSCLC
Keywords: Brain metastasis; Apatinib; Radiotherapy; NSCLC; Drive gene negative
MeSH Terms: conditions — Brain Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib combined with Radiotherapy (Experimental): Drugs: Apatinib Apatinib (500 mg/d) was given orally for one week before the brain radiotherapy, and then, continued to be administered at the same way during the brain radiotherapy period (3 weeks). It was given for another one week after the end of the brain radiotherapy.
  Radiotherapy: Intensity-modulated radiotherapy (IMRT).
  According to the patients KPS score, GPA score, the number and size of metastatic lesions can be selected:
  1. 37.5Gy/15 fractions of whole brain irradiation for multiple brain metastases were more than 5;
  2. The whole brain was irradiated with 37.5Gy/15 and simultaneous integrated boost dose of 52.5Gy/15 to patients with 1-5 metastatic lesions.
  Interventions: Drug: Apatinib
- Radiotherapy alone (No Intervention): Radiotherapy: Intensity-modulated radiotherapy (IMRT).
  According to the patients KPS score, GPA score, the number and size of metastatic lesions can be selected:
  1. 37.5Gy/15 fractions of whole brain irradiation for multiple brain metastases were more than 5;
  2. The whole brain was irradiated with 37.5Gy/15 and simultaneous integrated boost dose of 52.5Gy /15 to patients with 1-5 metastatic lesions.

INTERVENTIONS:
Drug: Apatinib — radiotherapy with Apatinib
  Other Names: Apatinib Mesylate
  Arms: Apatinib combined with Radiotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of concurrent radiotherapy with Apatinib in patients with Brain Metastases from drive gene wide-type Non-small-cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
Brain metastases (BM) develop in 22-54% of NSCLC patients during the disease course. NSCLC patients with BM with a median overall survival (OS) of 2-3 months when treated with systemic corticosteroid alone, and a median OS of 3-6 months when treated with whole brain radiation therapy (WBRT). Recently, several studies have reported the benefits of epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKIs) for EGFR mutation NSCLC patients with BM. The median OS of EGFR mutation patients with BM significantly improved with TKIs treatment, which ranged from 11.8 to 18.8 months. However, for the EGFR wide-type NSCLC patients with BM, the prognosis remains poor.

It was found that the combination of anti-VEGF drugs and brain radiotherapy can not only reduce the volume of peritumoral brain edema (PTBE), reduce the intracranial pressure, relieve the symptoms of nerve compression, reduce the risk of brain hernia during brain radiotherapy, and but also inhibit the hypoxia of tumor cells, increase the radiosensitivity of tumor cells, and ultimately improve the efficacy of radiotherapy.

Apatinib, a tyrosine kinase inhibitor that selectively inhibits the vascular endothelial growth factor receptor (VEGFR) and mildly inhibits c-Kit and c-SRC, has been reported to show efficacy among some patients with malignant supratentorial gliomas.

Therefore, the investigators initiated this study to evaluate the efficacy and safety of concurrent radiotherapy with Apatinib in patients with Brain Metastases from drive gene wide-type Non-small-cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, male or female, signed informed consent;
2. The primary lesion is confirmed by histopathology. The patient with brain metastases confirmed by histopathology or imaging confirmed the brain metastases. All patients with non-small cell lung cancer brain metastases should be recommended for EGFR mutation and ALK gene rearrangement assay，exclusion of patients with NSCLC brain metastases with positive EGFR-sensitive mutations and ALK gene rearrangement detection for TKI treatment; After multidisciplinary consultation and evaluation, patients with single or local multiple metastatic tumors with well-controlled primary lesions, who have the economic ability and are willing to undergo surgery for brain metastatic tumors were excluded.
3. Observable imaging data such as CT, MRI, etc., have measurable lesions as defined by RECIST 1.1 (R09-0262);
4. ECOG PS score: 0-2;
5. Hemogram index: RBC≥3.0×1012/L, WBC≥3.5×109/L, ANC≥1.5×109/L, PLT≥100×109/L, Hb≥90g/L
6. the expected survival time ≥ 3 months
7. Renal function: Cr≤1.2×UNL (upper limit of normal value);
8. Liver function: total bilirubin ≤ 1.5 × UNL; ALT, AST ≤ 1.5 × UNL

Exclusion Criteria:

1. . Allergies, known to be hypersensitive to any excipients in the study drug. ;
2. . Patients with recurrent brain metastases have previously received brain radiation therapy
3. . Patients with high fever and acute infection;
4. . Patients with active, progressive bleeding or a significant bleeding tendency in the primary lesion;
5. . Participated in any clinical trial of research drugs within 4 weeks prior to enrollment
6. . Diarrhea is the main symptom of the important or newly diagnosed acute gastrointestinal diseases, such as Crohn's disease, malabsorption or any cause of CTC ≥ 2 grade diarrhea.
7. . Current clinically relevant cardiovascular disease or medical history, such as refractory hypertension, NYHA grade 3 congestive heart failure, unstable angina or poorly controlled arrhythmias. Myocardial infarction occurred 6 months before randomization.
8. . Absolute neutrophil count <1000/mm3;
9. . Platelet count <50000/mm3;
10. . According to the investigator's point of view, any other serious disease or organ system dysfunction that may affect patient safety or interfere with the safety assessment of the test drug, such as proteinuria (CTCAE4.0-≥3), severe liver and kidney dysfunction (CTCAE4.0-≥3), hand-foot syndrome (CTCAE4.0-≥3) and so on.
11. . There are ulcers, intestinal perforations, and intestinal obstruction.
12. . Pregnant and lactating women
13. . Suspected or indeed have a history of alcohol and drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression-free survival (iPFS) | Evaluated in 24 months since the treatment began
  Defined as the time from randomisation to progression of intracranial disease or death from any cause.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 4 weeks after Radiotherapy.
  Proportion of patients with reduction or keeping in stable in tumor burden of a predefined amount
Objective response rate (ORR) | 4 weeks after Radiotherapy.
  Proportion of patients with reduction in tumor burden of a predefined amount
intracranial time to progress (ITTP) | Tumor assesment at 4 weeks and 12 weeks after radiotherapy, and then every 12 weeks, up to 24 months
  Defined as the time from randomisation to progression of intracranial disease
Overall survival (OS) | Tumor assesment at 4 weeks and 12 weeks after radiotherapy, and then every 12 weeks, up to 24 months
  Defined as the time from randomisation to death from any cause
Rate of Peritumoalbrainedema (PTBE) | 4 weeks after Radiotherapy.
  PTBE volume was measured in a similar manner by measuring the high SI region in T2WI that was clearly distinguished from normal tissues, including the tumor. Edema index was calculated by dividing the PTBE volume by tumor volume. The Edema index represents the degree of the PTBE, compared to tumor volume, with an index of 1.0 indicating no PTBE development.

CONTACTS AND LOCATIONS:
Overall Officials: Desheng Hu, Study Director — Associate dean
Locations (1):
- Hubei Cancer hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Ma J, Pi G, Bi J, Li Y, He H, Li Y, Hu D, Verma V, Han G. Concurrent Apatinib and Brain Radiotherapy in Patients With Brain Metastases From Driver Mutation-negative Non-small-cell Lung Cancer: Study Protocol for an Open-label Randomized Controlled Trial. Clin Lung Cancer. 2021 Mar;22(2):e211-e214. doi: 10.1016/j.cllc.2020.10.007. Epub 2020 Oct 21. PMID 33187916